CLINICAL TRIAL: NCT01835574
Title: Cambodia Integrated HIV and Drug Prevention Implementation Program
Acronym: CIPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1R01DA033672 (NIH)
Record Dates: First submitted 2013-04-09; First posted 2013-04-19 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: HIV
Keywords: Amphetamine-type substance use

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Conditional Cash Transfer and Cognitive-behavioral aftercare (Other): Pre- and post- CCT+AC intervention comparison
  Interventions: Behavioral: Conditional cash transfer and cognitive-behavioral aftercare

INTERVENTIONS:
Behavioral: Conditional cash transfer and cognitive-behavioral aftercare — The intervention combines a 12-week conditional cash transfer (CCT) intervention with 4-weeks of cognitive-behavioral group aftercare (AC) among women who use ATS. CCT includes thrice weekly urine screening for 12 weeks; participants receive $ for ATS-negative screens. Those with 3 negative screens in a week participants receive a cash bonus, which increase per month to mitigate habituation to the CCT reward schedule. Women who complete >=50% of ATS negative screening visits may participate in a 4-week, cognitive-behavioral AC group delivered immediately after CCT, which includes: 1) experiential group exercises; 2) didactic recovery skills training; 3) meditation and relaxation training; and 4) a ''lucky draw'' which is a form of CCT that provides positive reinforcement for group attendance.

SUMMARY:
HIV risk among female entertainment and sex workers (FESW) remains high and use of amphetamine-type stimulants (ATS) significantly increases this risk. We designed a cluster randomized stepped wedge trial: The Cambodia Integrated HIV and Drug Prevention Implementation [CIPI) study. The CIPI study is embedded within the SMARTgirl HIV prevention program. The CIPI study aimed to recruit FESW from 10 provinces, assessing HIV risk exposures including ATS use. The CIPI study then tested sequentially delivered, behavioral interventions targeting ATS use. The trial combines a 12-week Conditional Cash Transfer (CCT) intervention with four-weeks of cognitive-behavioral group aftercare (AC) among FESW who use ATS. The primary goal of the CIPI study is to reduce ATS use and unprotected sex among FESW. The CCT+AC intervention is being implemented in ten provinces where order of delivery was randomized. Outcome assessments (OEs) including biomarkers and self-reported measures of recent sexual and ATS use behaviors are conducted prior to implementation, and at three 6-month intervals after completion. All women who are ATS negative at 6-months, including those who have completed the CCT+AC intervention are eligible to participate in a micro-enterprise (ME) opportunity. Consultation with multiple groups and stakeholders on implementation factors facilitated acceptance and operationalization of the trial. Statistical power and sample size calculations were based on expected changes in ATS use and unprotected sex at the population level as well as within-subjects. Dissemination of process indicators during the multi-year trial is carried out through annual in-country Stakeholder Meetings. Provincial 'Close-Out' forums are held at the conclusion of data collection in each province. When analysis is completed, dissemination meetings will be held in Cambodia with stakeholders, including community-based discussions sessions, policy briefs, and results published and presented in the HIV prevention scientific journals and conferences. CIPI is the first trial of an intervention to reduce ATS use and HIV risk among FESW in Cambodia. Results will inform both CCT+AC implementation in low and middle-income countries and programs designed to reach FESW.

DETAILED DESCRIPTION:
The CIPI Study is 16-week program that combines Conditional Cash Transfer (CCT) and group-based supportive After Care (AC) for moderate and high risk FESW ATS users using a stepped wedge randomized cluster design. The trial tests the CCT+AC intervention in 10 Cambodian provinces (clusters). Outcome Evaluation (OE) data is collected at 1 time-point prior to implementation of the CCT+AC program (Baseline), and 3 time-points after the intervention (OE-1, OE-2, and Post-OE) at 6, 12, and 18 months after baseline in each province. CCT+AC is followed by a linked economic capacity building opportunity. Women who are ATS-free, including those negative at baseline and those who successfully complete the CCT+AC intervention are eligible for referral to a MicroEnterprise (ME) program. The ME program combines financial literacy education and referral to a Cambodian registered microfinance organization (Chamroeun) for loan applications that may support alternate economic options for participating eligible women.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* biological female
* speaks Khmer language
* self reports 2 or more sex partners and/or transactional sex in last month
* able to provide informed consent

Exclusion Criteria:

* male sex
* under 18 years of age
* unable to speak Khmer language
* unable to consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1198 (Actual)
Dates: Start 2013-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Sexual risk | 6, 12 and 18 months
  Change in number of sexual partners in the past 3 months (measured as a numeric variable).
Amphetamine type stimulant use (ATS) | 6, 12, and 18 months
  Change in ATS use as measured by urine toxicology screening.

SECONDARY OUTCOMES:
Sexual risk 2 | 6,12, and 18 months
  Number of new sexual partners in the past 3 months.
Sexual risk 3 | 6, 12 and 18 months
  Biomarker outcome (prostate specific antigen (PSA)) indicating unprotected vaginal sex Biomarker outcome (prostate specific antigen (PSA)) indicating unprotected vaginal sex
Sexual risk 4 | 6,12, and 18 months
  Condom use with all paying partners
Sexual risk 5 | 6,12, and 18 months
  Condom use with all non-paying partners
ATS 2 | 6,12 and 18 months
  Self-reported ATS use using ASSIST
ATS 3 | 6, 12, and 18 months
  Self-reported binge use of ATS

OTHER OUTCOMES:
Recent alcohol use | 6, 12, and 18 months
  Self-reported alcohol use as measured by ASSIST
Hazardous drinking | 6, 12, and 18 months
  Self-reported alcohol use as measured by AUDIT-C
HIV and STI service use | 6, 12 and 18 months
  HIV testing and STI diagnoses
Reproductive health outcomes | 6, 12 and 18 months
  (i) visits to reproductive health clinics, (ii) birth control use, (iii) pregnancy termination
Economic well being | 6,12, and 18 months
  (i) income, (ii) housing instability, (iii) food insecurity, (iv) number of electronic devices in the home
Psychological distress | 6, 12, and 18 months
  Kessler 10 scale score

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Page, PhD., Principal Investigator — University of New Mexico Health Sciences Center
Locations (1):
- Family Health International, Phnom Penh, Cambodia

IPD SHARING:
Plan to Share IPD: No
No plan to share individual level data at this time outside of study investigators.

REFERENCES:
- [Background] Page K, Stein ES, Carrico AW, Evans JL, Sokunny M, Nil E, Ngak S, Sophal C, McCulloch C, Maher L. Protocol of a cluster randomised stepped-wedge trial of behavioural interventions targeting amphetamine-type stimulant use and sexual risk among female entertainment and sex workers in Cambodia. BMJ Open. 2016 May 9;6(5):e010854. doi: 10.1136/bmjopen-2015-010854. PMID 27160844
- [Background] Carrico AW, Nil E, Sophal C, Stein E, Sokunny M, Yuthea N, Evans JL, Ngak S, Maher L, Page K. Behavioral interventions for Cambodian female entertainment and sex workers who use amphetamine-type stimulants. J Behav Med. 2016 Jun;39(3):502-10. doi: 10.1007/s10865-016-9713-2. Epub 2016 Jan 18. PMID 26782667
- [Background] Dixon TC, Ngak S, Stein E, Carrico A, Page K, Maher L. Pharmacology, physiology and performance: occupational drug use and HIV risk among female entertainment and sex workers in Cambodia. Harm Reduct J. 2015 Oct 16;12:33. doi: 10.1186/s12954-015-0068-8. PMID 26472570
- [Derived] Muth S, Len A, Evans JL, Phou M, Chhit S, Neak Y, Ngak S, Stein ES, Carrico AW, Maher L, Page K. HIV treatment cascade among female entertainment and sex workers in Cambodia: impact of amphetamine use and an HIV prevention program. Addict Sci Clin Pract. 2017 Sep 5;12(1):20. doi: 10.1186/s13722-017-0085-x. PMID 28870232